CLINICAL TRIAL: NCT06124235
Title: Assessment of Coated Orthodontic Miniscrews With Chlorhexidine Hexametaphosphate Antimicrobial Nanoparticles (A Randomized Clinical Trial)
Brief Title: Assessment of Coated Orthodontic Miniscrews With Chlorhexidine Hexametaphosphate Antimicrobial Nanoparticles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Ali Abbas, Bachelor's dental Surgery ( B. D. S), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Coated Orthodontic Miniscrews
Record Dates: First submitted 2023-10-19; First posted 2023-11-09 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Orthodontic Appliance Complication
Keywords: Orthodontic miniscrew; Success Rate; Miniscrew Mobility; Pain Perception; Peri-implant health; Coated miniscrew; Coated Mini-implant; Chlorhexidine Hexametaphosphate Antimicrobial Nanoparticles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coated Miniscrew (Experimental): Device Place stent for accurate position of miniscrew, x-ray, inserting miniscrew, xray for showing position of miniscrew, then use Visual analoge scale for pain assessment for first 7 days, peri-implant health and mobility check each month for 3 month and success rate after 4 month.
  Interventions: Combination Product: Coated Orthodontic Miniscrews with Chlorhexidine Hexametaphosphate Nanoparticles
- Uncoated Miniscrew (Active Comparator): Device Place stent for accurate position of miniscrew, x-ray, inserting miniscrew, xray for showing position of miniscrew, then use Visual analoge scale for pain assessment for first 7 days, peri-implant health and mobility check each month for 3 month and success rate after 4 month.
  Interventions: Combination Product: Uncoated Miniscrew with Chlorhexidine Hexametaphosphate Nanoparticles

INTERVENTIONS:
Combination Product: Coated Orthodontic Miniscrews with Chlorhexidine Hexametaphosphate Nanoparticles — insertion:
  1. According to the random number generated, the corresponding envelop for left and right side by chosen.
  2. The patient will be asked to brush his/her teeth.
  3. The patient will rinse his/her mouth with chlorhexidine mouth rinse (0.12%) just before surgery being at least half an hour after brushing.
  The miniscrews used conical shaped, self-drilling, 1.6 mm in diameter, 8mm in length made of Ti.
  1. The site of insertion determined from the x-ray by using stent that will be fabricated for accurate site for OMS.
  2. Infiltration LA will be administered. Approximately 0.45 mL ,injected into the alveolar mucosa above the OMS placement site, in order to provides an acceptable anesthesia, while still allowing the patient feedback in case the OMS contacting the periodontal ligament (PDL).
  3. OMS will be placed manually by screw driver on buccally at an angle 90 degrees and then adjusted to the appropriate angle.
  4. x-ray will be taken to confirm OMS position.
  Arms: Coated Miniscrew
Combination Product: Uncoated Miniscrew with Chlorhexidine Hexametaphosphate Nanoparticles — Non-coated orthodontic miniscrews
  Arms: Uncoated Miniscrew

SUMMARY:
Aim To compare between orthodontic miniscrews coated and uncoated with CHX- HMP NP nanoparticles.

DETAILED DESCRIPTION:
Anchorage management by using of OMS to give anchoring for force application made using several orthodontic treatment techniques simple and improved their efficacy , because anchorage control is a challenge throughout the orthodontic treatment process till temporary orthodontic anchorage devices have been developed. Although stainless steel (SS) screws were initially introduced, the majority of currently presented OMS are manufactured from titanium (purity grades I to IV). Because they offer greater mechanical strength and reduce the danger of fracture during insertion and removal, titanium alloy miniscrews are typically employed. Failure of these devices is the most frequent issue related to the usage of OMSs. The development of a biofilm on these devices that causes periimplantitis is one of the recognized reasons for failure.

Primary stability (mechanical stability) is awarded shortly after the placement procedure of the device and secondary stability (biological stability) initiates at the placement time and enhances during the process of healing or bone remodeling. The first 8 weeks after insertion, during which time the stability of the implant transitions from mechanical to biological stability, are when OMS failure occurs most frequently. Although failure might be prevented by following the right protocols of treatment, the fact that, rate of failure of OMS could not be overlooked. The miniscrew's mobility and displacement, together with an infection of the soft tissues around, are causes of failure. Unmodified titanium and its alloys are prone to bacterial infections which lead to inflammation and failure of the implant eventually. Prevention of bacterial adhesion may inhibit biofilm formation.

Antibiotics used for protection against implant infection postoperatively is debatable due to inducing the process of antimicrobial resistance, substitute techniques to avoid this must be inspected. There are three recent solutions that have the ability to prevent the formation of biofilm on miniimplant surfaces. These include altering the topography of surfaces to prevent bacterial adhesion, treating surfaces with antimicrobial releasing agents for a set period of time to prevent bacterial adhesion, as well as eliminating bacteria nearby, and, finally, coating surfaces with antimicrobial agents that prevent attachment of bacteria over an extended period of time. The previous study on human dermal fibroblast of neonate cells showed that both coated and uncoated titanium OMSs were non-cytotoxic, furthermore, the animal study showed enhanced bone-remodeling process.

The research question is 'Does coating orthodontic mini-screws with CHX-HMP NPs increase their success rate?

ELIGIBILITY:
Inclusion Criteria:

* Undergoing orthodontic treatment by fixed orthodontic appliance.
* Indicated for a bilateral miniscrews.
* Good oral hygiene.

Exclusion Criteria:

* Medically compromised patients.
* Heavy smoker.
* Dry mouth ( Xerostomia).
* mucogingival lesions.
* Patients with chlorhexidine allergy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Compare the success rate of coated and uncoated miniscrews. | for 4 month.
  Orthodontic mini-screw will be considered successful when it could be loaded with orthodontic forces and fulfill its anchorage objectives without pain, gingival growth cover the head of miniscrew and fracture of miniscrew.

SECONDARY OUTCOMES:
Comparing the peri-implant health around coated and uncoated miniscrews. | each month for 3 month.
  The absence versus presence of peri-implantitis was evaluated by means of periodontal visual inspection. When the keratinized gingiva were normal (i.e., they had a pink color, no edema or tissue growth, and no spontaneous bleeding), they were given a score of 0 (absence of peri-implantitis). A score of 1 was used to indicate mild peri-implantitis (i.e., the keratinized gingiva around the MI exhibited a color alteration, with a small volumetric increase, but not covering the MI head base, and without spontaneous bleeding. A score of 2 was used to indicate severe peri-implantitis, with the keratinized gingiva showing a color change, spontaneous bleeding, and gingival hyperplasia covering the MI head base. Finally, larger gingival hyperplasia covering part or all of the MI's head were given a score of 3. Normally, in the latter situation, the gingiva also presented with a color change and spontaneous bleeding.
Comparing pain perception between coated and uncoated miniscrews. | 1 day, 2 day, 3 day, 4 day, 5 day, 6 day, and 7 day.
  The patients will be given a sheet contain VAS scale and will be informed about how to use it. They will be told that zero in VAS corresponds to no pain and 10 corresponds to maximum pain, and will be asked to document their perceived pain intensity accordingly. Pain perception will be recorded after TAD insertion by 1 day, 2 day, 3 day, 4 day, 5 day, 6 day, and 7 day.
Comparing the miniscrew mobility between coated and uncoated miniscrews. | each month for 3 month.
  MI mobility was classified using 4 scores: a score of 0 was given when there was no movement of the MI. When there was a small amount of mobility of the MI, but without tissue ischemia, it was classified with score of 1 (exhibiting mobility but fulfilling its function). Moderate displacement of the MI causing tissue ischemia was classified with score of 2 (exhibiting displacement but fulfilling its function). Finally, a score of 3 was used when mobility was excessive, to the point of preventing the MI from maintaining anchorage.

CONTACTS AND LOCATIONS:
Overall Officials: Akram F. Alhuwaizi, Prof., Study Director — akramalhuwaizi@codental.uobaghdad.edu.iq
Locations (1):
- University of Baghdad College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
It will be mostly available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1/11/2024 If not affected on publishing of may article for 3 month can i share this information
Access Criteria: I can provide data as word or excel.

REFERENCES:
- [Derived] Al-Hilaly AA, Alhuwaizi AF. Assessment of coated orthodontic miniscrews with chlorhexidine hexametaphosphate antimicrobial nanoparticles: A randomized clinical trial. J World Fed Orthod. 2025 Apr;14(2):67-75. doi: 10.1016/j.ejwf.2024.09.006. Epub 2024 Nov 8. PMID 39521698